CLINICAL TRIAL: NCT04395443
Title: A Comparative Prospective Interventional Study Shows The Impact Of The Clinical Pharmacists' Role In The Emergency Department In Medication Reconciliation Upon Patients' Admission To Reduce The Medication Discrepancies.
Brief Title: The Impact Of Clinical Pharmacists Medication Reconciliation Upon Patients Admission To Reduce Medication Discrepancies.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alexandria University (Other)
Responsible Party: Principal Investigator, Heba Shaker, Supervisor of clinical pharmacy units in Alexandria Main University Hospital, Alexandria University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 0304494
Record Dates: First submitted 2020-05-16; First posted 2020-05-20 (Actual); Last update posted 2022-10-13 (Actual); Status verified 2020-12

CONDITIONS: Medication Reconcilitation Upon Hospital Admission
Keywords: Medication reconcilitation; Medication discrepancies; Admission pharmacist
MeSH Terms: interventions — Medication Reconciliation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- patients admitted to emergency department (Experimental): the intervention is the medication reconciliation
  Interventions: Other: medication reconciliation

INTERVENTIONS:
Other: medication reconciliation — the emergency clinical pharmacists will start medication reconciliation with the admitted patients and a full diseases and preadmission medications history will be taken.A comparison between the accuracy and completeness of drug history lists already presented in the profile and drug history taken by the clinical pharmacists to detect the medication discrepancies

SUMMARY:
It is a quazai one arm study shows the impact of the role of the clinical pharmacists through medication reconciliation to patients admitted to the emergency department .The main aim is to show if the pharmacists intervention is associated with establishing a complete drug history list than the list already presented in the patient file and taken by the physician .Then a description of the medication errors detected will be done .

DETAILED DESCRIPTION:
It is a quazai one arm study in which the pre phase is the detection of the complete and accurate drug history list already presented in the patient file and taken by the physician and the post phase is the detection of the complete and accurate drug history list taken by the clinical pharmacists after medication reconciliation for the same patients.

medication reconciliation will be done as a full diseases and preadmission medications history will be taken from the patients or the family through interviews, revising previous prescriptions and hospital records.

* Preadmission medication history will include medications trade names, doses, frequency and route of administration and treatment duration and also will include the consumption of vitamins or herbs.
* The medication errors will be detected ,calculated and classified according to medication at transitions and clinical handoffs (MATCH) toolkit for medication reconciliation and NCC MERP index.

ELIGIBILITY:
Inclusion Criteria:

* Patients with one or more chronic disease / drug.

Exclusion Criteria:

- Patients who cannot communicate or have no family members.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 161 (Actual)
Dates: Start 2020-09-25 (Actual); Primary Completion 2020-11-30 (Actual); Study Completion 2020-11-30 (Actual)

PRIMARY OUTCOMES:
the total number of complete and accurate drug history list detected in each phase. | 2 months
  to calculate the total number of complete and accurate drug history list taken by the physicians and already presented in the profile (pre phase) and the total number of complete and accurate drug history list taken by the clinical pharmacists after medication reconciliation (post phase).
Detect the number of medication discrepancies and the proportion of the prescriptions with one or more medication discrepancies | 2 months
  Calculate the total number of medication discrepancies detected after medication reconciliation and then calculate and the proportion of the prescriptions with one or more medication discrepancies from the total number of prescriptions.
  2- to classify the medication discrepancies using Medications at Transitions and Clinical Handoffs (MATCH) Toolkit for Medication Reconciliation.
  2- to classify the medication discrepancies using Medications at Transitions and Clinical Handoffs (MATCH) Toolkit for Medication Reconciliation.
  2- to classify the medication discrepancies using Medications at Transitions and Clinical Handoffs (MATCH) Toolkit for Medication Reconciliation.
  to classify the medication discrepancies using Medications at Transitions and Clinical Handoffs (MATCH) Toolkit for Medication Reconciliation and NCC MERP index
classification of medication discrepancies | 2 months
  to classify the medication discrepancies according to MATCH toolkit for medication reconciliation and NCC MERP index.
  3- to calculate the proportion of the patients detected with one or more medication discrepancies
  3- to calculate the proportion of the patients detected with one or more medication discrepancies
  3- to calculate the proportion of the patients detected with one or more medication discrepancies to calculate the proportion of the patients detected with one or more medication discrepancies
the total number of complete medication history lists will be written in the patients profiles | 2 months
  to calculate the total number of complete medication history lists will be written in the patients profiles by the clinical pharmacists after their interventions..

CONTACTS AND LOCATIONS:
Locations (1):
- Alexandria Main University Hospital, Alexandria, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Shaker HO, Sabry AAF, Salah A, Ragab GM, Sedik NA, Ali Z, Magdy D, Alkafafy AM. The impact of clinical pharmacists' medication reconciliation upon patients' admission to reduce medication discrepancies in the emergency department: a prospective quasi-interventional study. Int J Emerg Med. 2023 Dec 15;16(1):89. doi: 10.1186/s12245-023-00568-z. PMID 38102544

DOCUMENTS (1):
  • Study Protocol (2019-12-19): https://cdn.clinicaltrials.gov/large-docs/43/NCT04395443/Prot_000.pdf